CLINICAL TRIAL: NCT06432920
Title: A Wearable In-phase Chest Wall Vibration Device for Relief of Dyspnoea in COPD: a First-in-human Exploratory Study
Acronym: ResWave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elevre Medical Ltd. (Industry)
Collaborators: Beacon Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RW-CIP 1.2
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
Keywords: dyspnea; COPD; chronic obstructive pulmonary disease; cpet; cardiopulmonary exercise testing; chest wall vibration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Participants undergo constant-work rate cardiopulmonary exercise testing 2 times: once while wearing the active prototype device (intervention) and once wearing the inactive prototype device (control). Order of intervention/control is randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ResWave (Experimental): In-phase Chest Wall Vibration worn and active during constant work rate exercise testing.
  Interventions: Device: ResWave
- Control (Placebo Comparator): In-phase Chest Wall Vibration worn and inactive (off) during constant work rate exercise testing.
  Interventions: Device: ResWave

INTERVENTIONS:
Device: ResWave — Prototype wearable in-phase chest wall vibration device

SUMMARY:
The goal of this exploratory clinical trial is to evaluate the initial clinical safety and performance of a prototype wearable chest wall vibration (CWV) device intended to relieve exertional dyspnea in adults with Chronic Obstructive Pulmonary Disease. The main questions it aims to answer are:

* Can CWV be delivered safely to participants via a wearable device?
* Is there evidence of an effect on participant-reported dyspnea, endurance time and other measures of cardiorespiratory function?

Participants will undergo two cycle-ergometer exercise testing sessions while wearing the prototype wearable device. The device will be active in one session (intervention) and inactive in the other (control). The order in which intervention or control occurs will be randomised. Researchers gather data relating to adverse events, device deficiencies, participant-reported symptom severity, endurance time and measures of cardiorespiratory function recorded via standard CPET apparatus.

DETAILED DESCRIPTION:
The purpose of this Clinical Investigation is to evaluate the device design in a small number of human subjects with respect to initial clinical safety, and to gather preliminary data regarding the effect of the device on patient reported dyspnoea and physiological measures of cardiorespiratory function. This will facilitate planning of further steps of device development and validation, guide design modifications and define parameters for a future pivotal clinical investigation.

The investigational device is at Pilot stage of Clinical Development, and the proposed Clinical investigation is a first-in-human exploratory study. It is not a superiority, non-inferiority, or equivalence study.

The primary objective of this Clinical Investigation is to evaluate the investigational device with respect to initial clinical safety when used by subjects with Chronic Obstructive Pulmonary Disease during physical exertion in the form of cycle ergometer-based Cardiopulmonary Exercise Testing.

The secondary objective of this Clinical Investigation is to gather preliminary data regarding the effect of the device on patient-reported dyspnoea and physiological measures of cardiorespiratory function.

Each subject will attend the investigation site for a Pre-Study visit during which formal written consent will be obtained, clinical history and medications will be reviewed as part of standard CPET pre-assessment, and enrolment in the Clinical Investigation will be complete.

An initial Incremental Cardiopulmonary Exercise Testing (CPET) session will then be conducted to determine baseline Peak Work Rate capacity. This is necessary so that the intensity of CPET that will be required to achieve 75% of each subject's individual Peak Work Rate capacity can be determined. Peak Work Rate capacity will be defined as the highest work rate that the Subject is able to maintain for ≥30 seconds.

Following initial CPET, subjects will return for device testing on a non-consecutive day. Each subject will undergo 2 study arms during this visit: the Intervention (ResWave) and Control arms, in the random order. Both arms will be conducted on the same day, with a recovery period of 60 minutes between each arm. Subjects will undergo sub-maximal exercise testing at a Constant Work Rate (CWR) of 75% of their peak work rate capacity in both arms. Borg CR10 scores will be recorded at 2 minute intervals throughout. Endurance time will be recorded at test completion. Adverse Events will be recorded throughout testing and at 72-hour follow-up via phone call. Device Deficiencies will be recorded throughout testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) with FEV1 / FVC ratio of < 75% and deemed clinically stable
* Moderate to severe airflow limitation on Spirometry (FEV1: 30 to 75% predicted)
* Pulmonary Function Testing completed in the last 6 months

Exclusion Criteria:

* Active pulmonary infection or exacerbation within last 6 weeks
* Unstable cardiac disease - cardiac intervention, change in symptoms or medication within last 6 weeks
* BMI > 35
* Receiving domiciliary oxygen therapy
* Diagnosis of COVID-19 within the last 12 weeks or persistent symptoms directly attributable to previous COVID-19 infection
* Presence of comorbid condition that is deemed to be a significant contributor to dyspnoea: Heart Failure, Chronic Thromboembolic Disease, Neuromuscular Disease, Primary Pulmonary Hypertension
* Pulmonary Embolism in last 3 months
* Abdominal or Thoracic surgery in last 3 months
* Pneumothorax in last 6 months
* Active malignancy
* Active chest wall pain, active skin condition or open wound on thorax
* Pregnant or breastfeeding
* Women of child-bearing age (premenopausal, under age 50, or without previous sterilisation surgery)
* Any implantable electronic device
* On anticoagulants or with known history of coagulopathy
* Any absolute or relative contraindication to CPET testing
* Disability or comorbid condition that prevents exercise training and/or use of CPET apparatus and/or wearing the investigational device
* Previous experience of Chest Wall Vibration therapies for relief of breathlessness
* Currently enrolled in any other clinical trial or research study
* People deemed to be incapable of giving consent, or with reduced capacity to consent or diminished autonomy as a result of mental or cognitive impairment, or deemed otherwise vulnerable on clinical grounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 72 hours
  Adverse Events during or following use of the prototype device and/or exercise testing protocol
Device Deficiencies | During active use in exercise testing
  Performance data of the device during use

SECONDARY OUTCOMES:
Dyspnea severity | Recorded at 2 minute intervals during exercise testing. Outcome measure at isotime.
  Borg Category-Ratio scale (Borg CR10). Scale from 0 (lowest intensity, better) to 10 (maximal intensity, worse).
Endurance time | Duration of exercise testing
  Exercise testing endurance time
Reason for stopping | During exercise testing
  Whether participant stopped exercise testing due to dyspnea or other reason
Minute Ventilation (VE) | During exercise testing
  Minute Ventilation in millilitres/minute (mL/min)
Heart Rate (HR) | During exercise testing
  Heart rate in beats per minute (BPM)
Oxygen Pulse | During exercise testing
  Oxygen Pulse (VO2/HR) in millilitres/minute (mL/min)
Oxygen Consumption | During exercise testing
  Oxygen Consumption (VO2) in millilitres/minute (mL/min)
Carbon Dioxide Production | During exercise testing
  Carbon Dioxide Production (VCO2) in millilitres/minute (mL/min)
Work | During exercise testing
  Work (W) in watts
Tidal Volume (VT) | During exercise testing
  Tidal Volume in Litres (L) at body temperature and pressure saturated (BTPS)
Respiratory Quotient (RQ) | During exercise testing
  Respiratory Quotient (CO2 produced / O2 consumed; no unit as it is a ratio value)
End-tidal carbon dioxide tension (PETCO2) | During exercise testing
  End-tidal carbon dioxide tension (PETCO2) in millimetres of mercury (mmHg)
End-tidal oxygen tension (PETO2) | During exercise testing
  End-tidal oxygen tension (PETO2) in millimetres of mercury (mmHg)
Oxygen Saturation (SpO2) | During exercise testing
  Oxygen Saturation (SpO2) (%, percentage)
Respiratory Reserve | During exercise testing
  Respiratory Reserve in Litres
Expiration Time | During exercise testing
  Expiration Time in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Professor Seamus Linnane (MB BCh BAO FRCP FRCPI), Principal Investigator — Beacon Hospital
Locations (1):
- Beacon Hospital, Sandyford, Dublin 18, Ireland

IPD SHARING:
Plan to Share IPD: No
At present there is no plan to share individual participant data (IPD). As this is a novel medical device prototype currently undergoing development, IPD sharing could undermine future research and development activities relating proprietary aspects of the technology.